CLINICAL TRIAL: NCT01749722
Title: Safety and Efficacy of the NaviAid™ G-Eye System During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smart Medical Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: G-Eye 15502
Record Dates: First submitted 2012-11-11; First posted 2012-12-17 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Colorectal Cancer; Polyp; Adenoma
Keywords: Colorectal Cancer; Polyp; Adenoma; Detection Rate; Colonoscopy; NaviAid™ G-Eye procedure; NaviAid™ G-Eye system; G-Eye procedure; G-Eye system
MeSH Terms: conditions — Colorectal Neoplasms; Polyps; Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NaviAid™ G-Eye procedure (Experimental): NaviAid™ G-Eye procedure
  Interventions: Device: NaviAid™ G-Eye procedure

INTERVENTIONS:
Device: NaviAid™ G-Eye procedure — NaviAid™ G-Eye procedure

SUMMARY:
To evaluate the safety of using the NaviAid™ G-Eye system during Colonoscopy

DETAILED DESCRIPTION:
Colonoscopy is the gold-standard method for CRC screening, as it enables detection and real-time removal of pre-cancerous polyps during the examination. It is well known that lesions are missed during routine colonoscopy.5 major reasons can be detailed for missing polyps during colonoscopy: polyps that are hidden behind folds, polyps that are masked by the colon's topography and natural folds, shallow polyps, unscreened portions of the colon (due to incomplete colonoscopy) and endoscope slippage. The NaviAid™ G-Eye system presents a unique concept that overcomes all 5 items listed above, providing an overall solution to the two endoscopy key challenges of limited detection/treatment yield and limited operation range.

The G-Eye endoscope comprises a standard endoscope onto which a unique balloon is permanently integrated, at its bending section. The NaviAid™ G-Eye may be used for performing controlled withdrawal and endoscope stabilization.

A major attribute of the NaviAid™ G-Eye system controlled withdrawal technique of the endoscope, with the balloon moderately inflated is to expand and stretch the intestinal lumen during endoscope withdrawal.

This is a single-center, non randomized open-label study intended to evaluate the serious adverse events prevalence when using the NaviAid™ G-Eye system during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* The patient is undergoing colonoscopy for screening, for surveillance of previous colon polyp(s) or for diagnostic evaluation.
* The patient is 40-75 years old;
* The patient must understand and provide written informed consent for the procedure.

Exclusion Criteria:

* Subjects with inflammatory bowel disease;
* Subjects with a personal history of polyposis syndrome;
* Subjects with suspected colonic stricture potentially precluding complete colonoscopy;
* Subjects with active diverticulitis or toxic megacolon;
* Subjects with a history of radiation therapy to abdomen or pelvis;
* Pregnant or lactating female subjects;
* Subjects who are currently enrolled in another clinical investigation.
* Subjects with routine oral or parenteral use of anticoagulants
* Subjects with recent (within the last 3 mounts) coronary ischemia or CVA (stroke)
* Any patient condition deemed too risky for the study by the investigator

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Subjects will be followed during the study period (approximatly 3 hours) and follow up will be done within 48-72 hours following the procedure
  To evaluate the safety of using the NaviAid™ G-Eye system during Colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Gralnek, Prof., Principal Investigator — Elisha Hospital
Locations (1):
- Elisha Hospital, Haifa, Israel

REFERENCES:
- [Derived] Gralnek IM, Suissa A, Domanov S. Safety and efficacy of a novel balloon colonoscope: a prospective cohort study. Endoscopy. 2014 Oct;46(10):883-7. doi: 10.1055/s-0034-1377968. Epub 2014 Sep 16. PMID 25225962